Official Title: Fundus Finding and Thiol-Disulfide Homeostasis in Gestational Diabetes

ClinicalTrials.gov Identifier: NCT05958927

Document Date: April 13, 2023

## Statistical analysis

NCSS (Number Cruncher Statistical System) 2007 (Kaysville, Utah, USA) program will be used. While evaluating the study data, the distribution of the data will be evaluated with the Shapiro-Wilk Test, as well as the descriptive statistical methods (Mean, Standard Deviation, Median, Frequency, Ratio, Minimum, Maximum). Mann-Whitney U test will be used in comparisons of two groups that do not show normal distribution of quantitative data, and Student's t test will be used in case of normal distribution. Chi-square analysis will be used to determine the relationship between qualitative data. In order to determine the relationship between quantitative data, Pearson correlation analysis will be used in case of normal distribution and Spearman's correlation